CLINICAL TRIAL: NCT00620009
Title: The Measurement of Empathy and Its Efficacy in Psychotherapy
Acronym: EMPATHY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Bhaskar N. Sripada, MD / Associate Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2002-0381
Record Dates: First submitted 2008-02-11; First posted 2008-02-21 (Estimated); Last update posted 2008-02-21 (Estimated); Status verified 2008-02

CONDITIONS: Psychotherapeutic Processes; Transference (Psychology)
Keywords: Empathy; Feedback; Psychotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Therapists and patients record their estimates of the patient's Global Assessment of Functioning, but do not discuss these estimates in therapy sessions.
- Empathy Feedback (Experimental): Therapists and patients record their ratings of the patient's Global Assessment of Functioning and discuss these ratings.
  Interventions: Behavioral: Empathy Feedback

INTERVENTIONS:
Behavioral: Empathy Feedback — Discussion of empathy ratings between patients and therapists during psychotherapy sessions.
  Arms: Empathy Feedback

SUMMARY:
The purpose of the research is to: 1) to test whether psychotherapy including immediate feedback of empathy data is more efficacious than therapy without such an exchange of data, 2) to measure the degree of accuracy of therapist's empathy and its relationship to the patient's estimate of the therapist's empathy.

DETAILED DESCRIPTION:
Objective: To develop and evaluate a feedback method for measuring and increasing therapists' empathic accuracy and reducing empathic errors in psychotherapy. Method: Sixteen (16) patient-therapist pairs were randomly assigned to intervention and control groups. All patients rated their own functioning using the GAF (Global Assessment of Functioning) and predicted the accuracy with which their therapists would estimate their ratings. Therapists rated the patient's GAF, predicted the patients' ratings of their own GAFs, and rated their confidence in their own predictions. In the intervention condition, therapist and patients discussed the previous session's ratings for a few minutes of the therapy session. Results: Intervention therapists showed greater empathic accuracy relative to controls on our empathy measure (t(14) = 2.69, p < .01) and increased empathy over time on the Barrett-Lenard Empathy subscale (t(32) = 3.21, p < .01). We also found significant effects on errors related to perceived accuracy of therapist empathy. Patients in the control group were found to perceive their therapists to be either more or less accurate than was actually the case (over/under-idealization), but such biases were not as strong in the intervention group. Similarly, therapists in the control group were likely to over-estimate their own accuracy (over-confidence) to a greater extent than intervention therapists. Affective responses to the instrument were positive overall and did not differ by condition. Conclusion: Empathy feedback and feedback concerning degrees of patient idealization and therapist confidence may be effective in improving functioning as well as in increasing empathic accuracy in psychotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient psychotherapy at University of Illinois at Chicago
* Age 18-65

Exclusion Criteria:

* Psychosis
* Suicidality
* Organic Brain Disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2002-06; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Patient Global Assessment of Functioning | 20 psychotherapy sessions

SECONDARY OUTCOMES:
Barrett-Lenard Relationship Inventory | Every 5th session, 20 sessions of psychotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Bhaskar N. Sripada, M.D., Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States